CLINICAL TRIAL: NCT06240546
Title: A Phase I, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LPM6690176 Capsules in Patients With Advanced Solid Tumors.
Brief Title: First-in-Human Study of LPM6690176 in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY01024/CT-CHN-101
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 2 mg/m2 (Experimental): LPM6690176 capsules administered 2 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 4 mg/m2 (Experimental): LPM6690176 capsules administered 4 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 8 mg/m2 (Experimental): LPM6690176 capsules administered 8 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 16 mg/m2 (Experimental): LPM6690176 capsules administered 16 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 24 mg/m2 (Experimental): LPM6690176 capsules administered 24 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 36 mg/m2 (Experimental): LPM6690176 capsules administered 36 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176
- 48 mg/m2 (Experimental): LPM6690176 capsules administered 48 mg/m2 on day 1-5 (qd) every two weeks.
  Interventions: Drug: LPM6690176

INTERVENTIONS:
Drug: LPM6690176 — Administered orally
  Other Names: LY01024

SUMMARY:
This study is a phase 1, first-in-human, open-label, dose-escalation and dose-expansion study designed to evaluate the safety and tolerability, pharmacokinetics characteristics and preliminary anti-tumor activity of LPM6690176 capsules in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed informed consent;
2. Age 18 ~ 75 years, male or female;
3. Patients with histologically or cytologically confirmed advanced or metastatic unresectable solid tumors, who failed or intolerant to standard anti-tumor therapy or lack of standard therapy;
4. According to RECIST 1.1 criteria,

   * Dose escalation phase: patients with at least one non-measurable lesion;
   * Dose expansion phase: patients with at least one measurable lesion;
5. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1;
6. Life expectancy≥ 3 months;
7. Adequate bone marrow, liver, kidney, metabolism and coagulation function (blood transfusion, colony stimulating factors, albumin, and blood products are not allowed to use within 14 days before enrollment);
8. Negative pregnancy test within 7 days before first dose of study drug treatment in women of childbearing age. Female patients with childbearing potential were to use effective contraception during and for 6 months after the first dose of study drug treatment. Male patients (female partners with childbearing potential) should take effective contraceptive measures during study drug treatment and until 4 months after last dose of study drug administration.

Exclusion Criteria:

1. Patients who have not recovered from AEs caused by previous anti-tumor therapy to ≤ Grade 1 (assessed according to NCI-CTCAE 5.0 criteria, excluding alopecia and ≤ Grade 2 peripheral sensory neuropathy);
2. Pleural effusion, pericardial effusion, or ascites requiring medical intervention or frequent drainage within 1 month before signed informed consent decided by the investigator;
3. Symptomatic brain metastasis, history of spinal cord compression or leptomeningeal metastasis;
4. Concomitant Diseases:

   * Any of the following diseases within 6 months before the first dose of study treatment: myocardial infarction, unstable angina, coronary artery/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, and serious arrhythmia requiring treatment;
   * Patients who require long-term anticoagulant therapy or anti-platelet therapy or require long-term use of non-steroidal anti-inflammatory drugs;
   * Patients with uncontrolled hypertension, hypertensive crisis or history of hypertensive encephalopathy;
   * Patients with increased risk of gastrointestinal ulcer or gastrointestinal bleeding tendency or gastrointestinal perforation tendency;
   * Patients with known active colitis within 8 weeks prior to screening, or diarrhea ≥4 times in 24 hours;
   * Active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 2 weeks before the first dose of study drug treatment;
   * HBsAg (+) and HBV DNA≥ 1×103 or HCV (+) or HIV (+);
   * Patients who have undergone major surgical procedures 4 weeks before the first dose of study drug treatment, or have severe injury, or requiring elective major surgery during the study, or have unhealed wounds, ulcers or fractures;
   * Exclusion criterion specific to dose expansion phase: patients who have any malignancy within 5 years before the first dose of study treatment except for the specific cancer under investigation in this study (cured carcinoma in situ of the cervix, basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of breast ductal are eligible).
5. Prior Medications:

   * Patients who received anti-tumor therapy within 4 weeks before the first dose of study drug treatment;
   * Received LPM6690176 capsules or other PLK-1 inhibitors therapy before enrollment;
   * Received live attenuated vaccination within 4 weeks before signed informed consent;
   * Use of strong inducers or strong inhibitors of CYP3A4 within 2 weeks or 5 half-lives of the medication before the first dose of study drug treatment;
   * Use of medications mainly metabolized by CYP2B6 within 2 weeks or 5 half-lives (which takes longer time) of the medication before the first dose of study drug treatment;
6. Patients who may receive other systemic anti-tumor therapy or local radical therapy of target lesions/non-target lesions during the study;
7. History of drug abuse, drug addiction, or alcoholism;
8. Known hypersensitivity to any component of the study drug;
9. Patients who participated in other clinical trials and received treatment within 1 month;
10. Pregnant or lactating women;
11. Other conditions that may elevate the risk of the patient or interfere the study results decided by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of dose-limiting toxicities (DLTs) | From the first dose of study drug treatment through Cycle 1 (28 days)
maximum tolerated dose (MTD) of LPM6690176 | From the first dose of study drug treatment through Cycle 1 (28 days)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Approximately 2 years
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Duration of response (DOR) | Approximately 2 years
  DOR is defined as the time from the first determination of an objective response (CR or PR) per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first, as assessed by the investigator
isease control rate (DCR) | Approximately 2 years
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease (SD) per RECIST v1.1 as assessed by the investigato
Progression-free survival (PFS) | Approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug treatment to the date of the first documentation of progressive disease or death, whichever occurs first, as assessed by the investigator using RECIST v1.1.
Overall survival (OS) | Approximately 3 years
  OS is defined as the time from the date of the first dose of study drug treatment to the date of death (due to any reason) or documented last contact
Maximum plasma concentration | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2 (28 days).
  Maximum plasma concentration (Cmax) of LPM6690176 and its N-demethylated metabolite after a single dose and multiple dose
Time to maximum plasma concentration | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2 (28 days).
  Time to maximum plasma concentration (Tmax) of LPM6690176 and its N-demethylated metabolite after a single dose and multiple dose.
Area under the plasma concentration-time curve | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2 (28 days).
  Area under the concentration versus time curve from time zero to the last quantifiable time point (AUClast) of LPM6690176 and its N-demethylated metabolite after a single dose and multiple dose; Area under the concentration versus time curve from time 0 extrapolated to infinite time (AUCinf) of LPM6690176 and its N-demethylated metabolite after a single dose and multiple dose.
Elimination half-life | From Pre-dose of Cycle 1 and up to Pre-dose of Cycle 2 (28 days).
  Elimination half-life (t1/2) of LPM6690176 and its N-demethylated metabolite after a single dose and multiple dose.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No